CLINICAL TRIAL: NCT05826782
Title: Kocaeli University
Brief Title: Effect of Antioxidant Food Supplement on Sperm Proteomic Structure and Semen Parameters
Acronym: Asthenospermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Collaborators: ECZACIBAŞI (Unknown)
Responsible Party: Principal Investigator, Naci Burak Cinar, MD, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 344119007
Record Dates: First submitted 2023-03-23; First posted 2023-04-24 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Asthenozoospermia
Keywords: infertility; antioxidant; proteomics
MeSH Terms: conditions — Asthenozoospermia; Infertility

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Active Comparator): The treated group
  Interventions: Biological: Proxeed Plus 2*1 A arm
- B (Placebo Comparator): The placebo group
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Proxeed Plus 2*1 A arm — Proxeed plus 2 x daily sachets (2*1) three mounths
  Arms: A
Biological: Placebo — Placebo 2 x daily sachets (2*1) three mounths
  Arms: B

SUMMARY:
Infertility is defined as the inability to become pregnant despite 12 months of regular and unprotected intercourse. Male factors include defects in sperm concentration, morphology and motility, among which low sperm motility (asthenozoospermia) is one of the most common types of male infertility and affects approximately 40% of all cases.

It has become clear that protein defects in spermatozoa and semen can cause fertilization failure by affecting sperm motility, and it is necessary to define proteins and related pathways precisely because they have an important role in the treatment phase.

Increasing evidence shows that free oxygen radicals that occur as a result of oxidative stress (OS) play a very important role in the etiology of male infertility.

A systematic review including 29 studies (19 randomized clinical trials and 10 prospective studies) examined the effect of antioxidant food supplementation and reported a positive effect on baseline semen parameters, advanced sperm function, outcomes of assisted reproductive therapy, and live birth rate.

Conversely, few studies have failed to confirm any positive effect of antioxidant therapy and even report a negative effect on male fertility. Therefore, there is no clear consensus on the clinical efficacy of antioxidant therapy yet.

Since the pathogenesis has not yet been clearly demonstrated, treatments are not based on evidence, but based on clinical experience.

Our aim was to randomly divide infertile male patients who applied to our clinic with the complaint of infertility and found asthenozoospermia (restricted sperm motility) in their semen analysis into two arms and examine the effects of antioxidant food supplementation on sperm motility and proteomic structure with a placebo-comparative, prospective, double-blind study (LC-MS/MS). analysis) is to reveal the metabolic pathways that may lead to restriction of movement. The effect of antioxidant food support on sperm parameters and free oxygen radical levels in the control spermiogram after 3 (three) months of treatment to be given to the patients will be measured by ELISA method and compared with pre-treatment values.

ELIGIBILITY:
Inclusion Criteria:

1. Being in the age range of 20-40
2. Be infertile ( 12 months intercourse without any contraception)
3. Due to infertility, you should apply to us and have a spermiogram detection of asthenozoospermia
4. Patients whose spouses have normal gynecological examinations
5. Patients with normal physical examinations
6. Patients with normal hormonal values (FSH, LH,PRL,Testosterone,Estrogen) -

Exclusion Criteria:

1. previous treatment for infertility
2. Previously due to infertility or for any reason take antioxidant food supplements
3. Surgery or physical examination due to varicocele detection of varicocele
4. Detection of endocrine disorder (Defect in serum blends)
5. Smokers and alcohol addiction
6. Detection of infection in the genital tract
7. Having a chronic illness -

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
sperm motility (%) | 12 weeks
  semen analysis (microscopic analysis)

SECONDARY OUTCOMES:
Proteomics analysis | 8 weeks
  Water for chromatography (LC-MS Grade)
oxidative stress | 4 weeks
  ROS (Human SOD1(Superoxide Dismutase 1, Soluble) ELISA)

CONTACTS AND LOCATIONS:
Locations (1):
- Naci Burak Çinar, Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No